CLINICAL TRIAL: NCT05600270
Title: Comparison Between an Angled-tip and Straight-tip Guidewire in Biliary Cannulation: a Prospective, Randomized Trial
Brief Title: Angled-tip vs. Straight-tip Guidewire in Biliary Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neev Mehta (Other)
Responsible Party: Sponsor-Investigator, Neev Mehta, Study Coordinator, Lahey Clinic
Organization: Lahey Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20223146
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Bile Duct Diseases
Keywords: ERCP
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Single-Blinded Trial
Who Masked: Participant
Masking Description: Single-blinded study with masking of participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Angled wire (Active Comparator): Angled guidewire intervention arm
  Interventions: Device: Angled guidewire
- Straight wire (Active Comparator): Straight guidewire intervention arm
  Interventions: Device: Straight guidewire

INTERVENTIONS:
Device: Angled guidewire — Cannulation of the common bile duct using an angled-tip guidewire during ERCP
  Arms: Angled wire
Device: Straight guidewire — Cannulation of the common bile duct using an straight-tip guidewire during ERCP
  Arms: Straight wire

SUMMARY:
The investigators aim is to compare outcomes between an angled-tip guidewire and a straight-tip guidewire in cannulation of the common bile duct during ERCP. This is a randomized, controlled, single-blinded study. The primary outcome is success of cannulation and secondary outcomes are incidence of post-ERCP pancreatitis, procedure duration, and rate of complication between the angled wire and straight wire.

DETAILED DESCRIPTION:
Wire-guided cannulation of the common bile duct is a standard technique utilized during Endoscopic Retrograde Cholangio-Pancreatography (ERCP) to ensure safe and effective access to the common bile duct via the ampulla of Vater. Due to the anatomy of the ampulla, and the orientation of the biliary orifice, a guidewire with an angled tip may allow easier and safer access to the common bile duct without inadvertent manipulation of the pancreatic duct. The investigators aim to assess the technical and clinical outcomes between an angled-tip guidewire (GW) compared to a straight-tip guidewire in wire-guided cannulation of the common bile duct. The investigators hypothesize that an angled-tip GW is associated with increased rate of successful cannulation, decreased procedure time and decreased rate of post-ERCP pancreatitis in wire-guided biliary cannulation during ERCP.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ERCP for cholangiography, bile or tissue sampling from the gallbladder or bile duct
* patients undergoing ERCP for treatment of biliary diseases (removal of common bile duct stones, biliary stent placement)

Exclusion Criteria:

* Patients who are less than 18 years old
* Pregnant patients
* Patients who have undergone previous bile duct cannulation or sphincterotomy
* Patients who have undergone prior endoscopic balloon dilation or needle-knife fistulotomy
* Patients who have undergone gastric surgery (Billroth gastrectomy II, Roux-en-Y gastric bypass)
* Patients with acute pancreatitis
* Patients who refuse endoscopic intervention
* Patients with ampullary tumor, duodenal stenosis, or pre-operatively proven pancreaticobiliary malunion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Joyce, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vihervaara H, Gronroos JM, Koivisto M, Gullichsen R, Salminen P. Angled- or straight-tipped hydrophilic guidewire in biliary cannulation: a prospective, randomized, controlled trial. Surg Endosc. 2013 Apr;27(4):1281-6. doi: 10.1007/s00464-012-2596-6. Epub 2012 Dec 19. PMID 23250671

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Angled Wire | Straight Wire
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Angled Wire | Straight Wire | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Full Range); unit: years] | 70.42 [33 to 93] | 60.66 [31 to 96] | 68.18 [31 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 21 | 16 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cannulation
Description: Rate of successful cannulation of common bile duct
Time Frame: Day of Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Angled Wire | Straight Wire
Number analyzed (Participants) | 33 | 33
Participants | 30 | 31

2. Secondary Outcome: Post ERCP Pancreatitis
Description: Number of participants who develop post ERCP pancreatitis
Time Frame: Procedure day and up to day 5 post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Angled Wire | Straight Wire
Number analyzed (Participants) | 33 | 33
Participants | 1 | 2

3. Secondary Outcome: Duration
Description: Total duration of procedure
Time Frame: Day of procedure
Measure: Mean (Full Range); unit: seconds
Arm/Group | Angled Wire | Straight Wire
Number analyzed (Participants) | 33 | 33
seconds | 1964.26 [557 to 8520] | 1569.03 [711 to 4368]

ADVERSE EVENTS:
Time Frame: Randomization on day of procedure to post procedure day 5
Arm/Group | Angled Wire | Straight Wire
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angled Wire (N=33) | Straight Wire (N=33)
Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0)
Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0)
Post ERCP Cholangitis (Infections and infestations) | 0 (0) | 0 (0)
post ERCP Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT05600270/Prot_SAP_000.pdf